CLINICAL TRIAL: NCT05886439
Title: A Study of LK101 Combined With PD-1 or PD-L1 Monoclonal Antibody in the Treatment of Lung Cancer to Evaluate the Safety, Tolerability and Preliminary Efficacy
Brief Title: LK101 Combined With PD-1 or PD-L1 Monoclonal Antibody in the Treatment of Lung Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jie Wang, Chief of Medical oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LK101-IIT02
Record Dates: First submitted 2023-05-06; First posted 2023-06-02 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — pembrolizumab; durvalumab; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LK101 injection combined with pembrolizumab (Experimental): patients with locally advanced or metastastic (stage IIIB-IV) NSCLC and received ≤3 lines systemtic therapy. eligible subjects will receive LK101 injection and pembrolizumab treatment.
  Interventions: Drug: LK101 injection (personlized neoantigen pulsed DC vaccine ); Drug: Pembrolizumab
- LK101 injection combined with durvalumab (Experimental): patients with extensive SCLC who failed with at least first-line standard therapy. eligible subjects will receive LK101 injection and durvalumab treatment.
  Interventions: Drug: LK101 injection (personlized neoantigen pulsed DC vaccine ); Drug: Durvalumab
- LK101 injection combined with Tislelizumab (Experimental): Eligible subjects will receive LK101 injection and tislelizumab treatment.
  Interventions: Drug: LK101 injection (personlized neoantigen pulsed DC vaccine ); Drug: Tislelizumab

INTERVENTIONS:
Drug: LK101 injection (personlized neoantigen pulsed DC vaccine ) — LK101 will be administered in a prime-boost schedule of 4 priming vaccination followed by 3 booster vaccinations.
Drug: Pembrolizumab — Patients will receive pembrolizumab(200mg IV) Q3W until disease progression (PD), intolerable toxicity.
  Arms: LK101 injection combined with pembrolizumab
Drug: Durvalumab — Patients will receive durvalumab (1500mg IV) Q3W until disease progression (PD), intolerable toxicity.
  Arms: LK101 injection combined with durvalumab
Drug: Tislelizumab — 200 mg administered once every 3 weeks (Q3W) via intravenous infusion, with each infusion lasting longer than 30 minutes.
  Arms: LK101 injection combined with Tislelizumab

SUMMARY:
This is a open lable, single-center phase Ib/IIa study for patients with local advanced or metastastic NSCLC or ES-SCLC, who failed with previous anti-PD-1/PD-L1 therapy (cohort 1 and cohort 2) and for patients with ocal advanced or metastastic NSCLC received the first line treatment (cohort 3). The aim is to observe and evaluate the safety, tolerability and efficacy of LK101 injection combined with pembrolizumab, durvalumab or tislelizumab respectively in the incurable NSCLC and SCLC.

DETAILED DESCRIPTION:
This study is designed to evaluate the safety and efficacy of LK101 injection combined with pembrolizumab or durvalumab, which devided into 3 cohorts:

cohort 1: patients with locally advanced or metastastic (stage IIIB-IV) NSCLC who has progressed/relapsed after anti-PD-1/PD-L1 therapy. eligible subjects will receive LK101 injection and pembrolizumab treatment.

cohort 2: patients with extensive SCLC who failed with at least first-line standard therapy with PD-L1. eligible subjects will receive LK101 injection and durvalumab treatment.

cohort 3: patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) with no driver gene mutation and PD-L1 expression and have not experienced disease progression after receiving chemotherapy combined with an anti-PD-1 therapy.

LK101 will be administered in a prime-boost schedule of 4 priming vaccination followed by 3 booster vaccinations. For the priming phase: LK101 administered once a week at Days 1, 8, 15, 22. For the booster phase: total of 3 vaccinations will be given, Q3W from the end of priming dose. Treatment can be continued according to the investigator's evaluation, subsequent treatment is administered Q6W.

Patients will receive a combination of pembrolizumab(200mg IV) Q3W in cohort 1, durvalumab (1500mg IV) Q3W in cohort 2, tislelizumab (200mg) Q3W, respectively, until disease progression (PD), intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent;
* ≥18years, male or female;
* cohort1: Histologically/cytologically confirmed locally advanced or metastastic Non-small lung carcinoma (NSCLC), and received systemic treatment for recurrence/metastasis ≤3 lines; cohort2: Histologically/cytologically confirmed extensive small-cell lung carcinoma (ES-SCLC); Cohort 1 and Cohort 2 required patients progressed/recurrenced after anti-PD-1/PD-L1treatment;
* Cohort 3: Histologically/cytologically confirmed locally advanced or metastatic non-small cell lung cancer (NSCLC) with no driver gene mutation and have PD-L1 expression, and who have not experienced disease progression after receiving chemotherapy combined with an anti-PD-1 therapy.
* Life expectancy of more than 3 months;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1;
* At least one measurable lesion according to RECIST 1.1;
* The sequencing of tumor were qualified;
* According to the invistigators' judgment, venous vascular conditions can meet the needs of apheresis;
* For adequate organ function, the patients need to meet the following laboratory indexes:

  * hematologic functions(No blood transfusion or treatment with blood components and without granulocyte colony stimulating factor in the past 14 days.):

    * the absolute value of neutrophils (ANC) ≥ 1.5x109/L;
    * the platelet count was ≥ 90x109/L;
    * the hemoglobin > 9g/dL;
  * Hepatic functions:

    * Total bilirubin ≤ 1.5 × normal upper limit (ULN); patients with liver metastasis allow ≤ 3 × ULN;
    * aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN (patients with liver metastasis allow ALT or AST ≤ 5 × ULN);
  * renal

    * Serum creatinine ≤ 1.5 × ULN and creatinine clearance (calculated by Cockcroft-Gault formula) ≥ 50ml;
    * patients with urinary protein ≥ + + and confirmed 24-hour urinary protein quantity > 1.0g;
  * Coagulation function is good, defined as international standardized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN;
  * Normal thyroid function is defined as thyroid stimulating hormone (TSH) within the normal range. If the baseline TSH is beyond the normal range, subjects with total T3 (or FT3) and FT4 within the normal range can also be enrolled;
* FBG of patients without type 2 diabetes ≤ 126 mg/dL or ≤ 7.0 mmol/L, and that of patients with type 2 diabetes ≤ 167 mg/dL or ≤ 9.3 mmol/L; Or glycosylated hemoglobin (HbA1c) ≤8%;
* If there is a risk of pregnancy, all patient (male or female) are required to take appropriate methods for contraception during the study until the 6th month post the last administration of study drug;
* Well compliance, cooperate with follow-up;

Exclusion Criteria:

* History of hypersensitivity reaction to any vaccine and/or anti-PD-1/PD-L1 formulation ingredients; Or have had a previous severe allergic reaction to other monoclonal antibodies; Subjects who had previously discontinued anti-PD-1 /PD-L1 therapy due to "infusion reaction" or immune-related AE;
* Patients who have received therapeutic tumor vaccine products (including peptide vaccine, mRNA vaccine, DC vaccine, etc.);
* Diagnosis of malignant diseases other than study disease within 5 years before screening (except for malignant tumors that can be expected to recover after treatment);
* Patients received systemic antitumor treatment within 2 weeks before the apheresis, or receive reasearch drugs or device therapy;
* Received radiotherapy within 2 weeks prior to screening;
* Toxicity caused by previous treatment did not recover to CTCAE (version 5.0) Grade 1 or below (except hair loss and peripheral neuropathy);
* The tumor compresses the surrounding important organs or the superior vena cava, or invades the mediastinal great blood vessels, the heart, .etc;
* Patients who have recewived allogeneic hematopoietic stem cell transplantation or organ transplantation;
* A history of medical conditions that may trigger seizures (requiring treatment with antiepileptic medications);
* Patients who have active brain metastases or cancerous meningitis. Patients with treated brain metastases are eligible if they have been treated with brain metastases, and clinically stable for atleast 3 months, no evidence of disease progression 4 weeks before. All neurological symptoms had recovered, and off steroids at least 7 days prior to screening;
* Diaginosied or suspected of having an active autoimmune disease;
* patients with poorly controlled pleural effusion, pericardial effusion, or ascites requiring repeated drainage, or received pleural effusion or ascites treatment within the past 3 months;
* History of significant cardiovascular and cerebrovascular disease occurred in the 6 months prior to screening,Any of the following cardiac criteria:

  * Mean resting corrected QT interval (QTc) > 470 ms;
  * Left ventricular ejection fraction (LVEF) ≤ 50%;
  * American New York heart association (NYHA) heart function ≥ 2 or higher;
  * serious arrhythmia;
  * poorly controlled hypertension;
  * other serious heart disease;
* Patients with interstitial pneumonia, except those inactive and do not require hormone therapy disease;
* Patients diagnosed with active infections that are poorly controlled by systemic treatment;
* Any of the following test results are positive: human immunodeficiency virus (HIV) antibody, treponema pallidum antibody, hepatitis C virus (HCV) antibody, hepatitis B virus (HBV) surface antigen (HBsAg), HBV DNA and novel coronavirus nucleic acid;
* Active tuberculosis (TB) during screening;
* Treatment with systemic steroids or other immunosuppressive agents within 14 days prior to screening;
* Vaccination within 4 weeks prior to screening;
* Major injuries and/or surgery =< 4 weeks prior to screening;
* Persons with a history of psychotropic substance abuse and inability to abstain or with a history of mental disorders;
* Pregnant or lactating women;
* Skin diseases, such as psoriasis, may prevent intradermal vaccines from reaching the target area;
* Other conditions regimented at investigators' discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
DLT | Continuously throughout the study until 90 days after Termination of the treatment
  incidence of Dose limited toxicity(DLT),incidence and severity of adverse events (AEs), serious adverse events (SAEs), and immune-related adverse events (irAEs); Clinically significant abnormal changes in laboratory tests and other tests.
AE | Continuously throughout the study until 90 days after Termination of the treatment
  incidence and severity of adverse events
irAE | Continuously throughout the study until 90 days after Termination of the treatment
  incidence and severity of immune-related adverse events
SAE | Continuously throughout the study until 90 days after Termination of the treatment
  incidence and severity of serious adverse events

SECONDARY OUTCOMES:
ORR | accessed up to 24 months from baseline
  Objective Response Rate (ORR)according to mRECIST 1.1 standard
DoR | 24 months
  Duration of remission
DCR | 24 months
  Disease Control Rate
TTR | 24 months
  Time to remission
TTP | 24 months
  Time to progression
PFS | 24 months
  Progression Free Survival
OS | 24 months
  Overall Survival
Immune response evaluation | 24 months
  T cell response, cytokines, etc.

OTHER OUTCOMES:
Tumor immune microenvironment before and after treatment | 24 months
  CD8+T cell, PD-1, PD-L1, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Wang, MD,PhD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No